CLINICAL TRIAL: NCT03399864
Title: Effectiveness of Musical Training in Reducing Depressive Symptoms, Enhancing Self-esteem and Quality of Life Among Hong Kong Chinese Childhood Brain Tumor Survivors - A Pilot Randomized Controlled Trial
Brief Title: Effectiveness of Musical Training in Hong Kong Chinese Childhood Brain Tumor Survivors
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The University of Hong Kong (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: UW16-023_2
Record Dates: First submitted 2018-01-08; First posted 2018-01-16 (Actual); Last update posted 2019-06-12 (Actual); Status verified 2019-06

CONDITIONS: Brain Neoplasms; Child
MeSH Terms: conditions — Brain Neoplasms

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental group (Experimental): Apart from receiving scheduled medical follow-up, the subjects in the experimental group will receive a weekly 45-minute lesson on musical training for 52 weeks. The musical training will be conducted by the Music Children Foundation and be implemented in a ratio of one subject to one qualified orchestral performer at the subjects' homes. A musical instrument will be assigned to each subject based on their interests and the results of the prior assessment of subjects' expiratory function and fine motor skills. The musical training will start at the lowest level, such as hitting simple notes and end at the highest level, such as playing an entire song.
  Interventions: Behavioral: musical training
- Control group (Other): The subjects will receive usual care, such as medical follow-up according to the schedule of the oncology units.
  Interventions: Other: usual care

INTERVENTIONS:
Behavioral: musical training — The subjects in the experimental group will receive weekly 45-minute lessons on musical training for 52 weeks.
  Arms: Experimental group
Other: usual care — The subjects in the control group will receive usual care, such as medical follow-up according to the schedule of the oncology units.
  Arms: Control group

SUMMARY:
This study aims to work out the effectiveness (effect size) of the musical training intervention in reducing depressive symptoms, improving self-esteem and quality of life among childhood brain tumour survivors and to examine the feasibility, appropriateness, and acceptability of implementing musical training intervention in clinical practice. Subjects in the experimental group will receive weekly 45-minute lessons on musical training for one year (52 weeks), while those in the control group will receive usual care.

DETAILED DESCRIPTION:
Musical training has been increasingly implemented to promote one's psychological well-being and cognitive functioning. For instance, to reduce depression, anxiety in psychiatric patients, to improve self-esteem and mood recognition in hospitalized adolescent patients diagnosed with "adjustment reaction to adolescence", to improve social skills of children with autism, to enhance reading skills and academic achievement in young poor readers, and to facilitate children's cognitive development. Nevertheless, the effectiveness of musical training in promoting psychological well-being, particularly to reduce their depressive symptoms and enhance self-esteem, and enhancing quality of life among the childhood brain tumour survivors is remain underexplored. It is of paramount importance to examine the effectiveness of musical training so as to ameliorate adverse disease- and treatment-related late effects, such as depression and low self-esteem, hence enhancing childhood brain tumour survivors' quality of life.

ELIGIBILITY:
Inclusion Criteria:

* Hong Kong Chinese children surviving from brain tumours with the Modified Mini-Mental Scale (MMSE) score of 18 or above
* be aged between 7 and 16 years
* able to speak Cantonese and read Chinese
* have completed treatment for at least two months
* have residual function of the upper extremities (i.e. be able to move the extremities, such as the fingers and arms, without assistance)

Exclusion Criteria:

* children who have undertaken any musical training following their cancer diagnosis
* survivors with evidence of recurrence or second malignancies
* survivors receiving palliative care

Ages: 7 Years to 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 60 (Actual)
Dates: Start 2017-02-20 (Actual); Primary Completion 2018-06-30 (Actual); Study Completion 2018-06-30 (Actual)

PRIMARY OUTCOMES:
Change in depressive symptoms from baseline at 12-month follow-up between intervention and control group. | 12-month follow-up
  The subjects' depressive symptoms will be assessed at 12-month after starting the intervention using the Chinese version of the Center for Epidemiological Studies Depression Scale for Children (CES-DC).
  The CES-DC is a commonly used tool in assessing the number of depressive symptoms of children and adolescent (Radloff, 1977). It consists of 20 items which are rated on a 4-point Likert scale from 0 to 3 (0= "not at all", 1 = "a little", 2 = "sometimes", 3= "a lot") regarding the subjects' feelings and experiences of last week. A possible scores ranging from 0 to 60 will be obtained after summing up all the items. Higher scores indicate greater number of depressive symptoms experienced. The cut-off score of this scale is 16, which indicates the children or the adolescents are currently experiencing a significant level of depressive symptoms.

SECONDARY OUTCOMES:
Depressive symptoms at baseline between intervention and control group | baseline
  Subjects' depressive symptoms will be assessed at baseline using the Center for Epidemiological Studies Depression Scale for Children (CES-DC).
  The CES-DC is a commonly used tool in assessing the number of depressive symptoms of children and adolescent. It consists of 20 items which are rated on a 4-point Likert scale from 0 to 3 (0= "not at all", 1 = "a little", 2 = "sometimes", 3= "a lot") regarding the subjects' feelings and experiences of last week. A possible scores ranging from 0 to 60 will be obtained after summing up all the items. Higher scores indicate greater number of depressive symptoms experienced. The cut-off score of this scale is 16, which indicates the children or the adolescents are currently experiencing a significant level of depressive symptoms. Subjects will be asked to respond to the Chinese version of the CES-DC at baseline.
Change in depressive symptoms from baseline at 6-month follow-up between intervention and control group | 6-month follow-up
  Change in depressive symptoms will be assessed at 6-month after starting the intervention using the Center for Epidemiological Studies Depression Scale for Children (CES-DC).
  The CES-DC is a commonly used tool in assessing the number of depressive symptoms of children and adolescent. It consists of 20 items which are rated on a 4-point Likert scale from 0 to 3 (0= "not at all", 1 = "a little", 2 = "sometimes", 3= "a lot") regarding the subjects' feelings and experiences of last week. A possible scores ranging from 0 to 60 will be obtained after summing up all the items. Higher scores indicate greater number of depressive symptoms experienced. The cut-off score of this scale is 16, which indicates the children or the adolescents are currently experiencing a significant level of depressive symptoms. Subjects will be asked to respond to the Chinese version of the CES-DC at 6-month after starting the intervention.
Level of self-esteem at baseline between intervention and control group | baseline
  The subjects' self-esteem will be assessed at baseline, using the Chinese version of the Rosenberg Self-Esteem Scale (RSES).
  The RSES is a tool designed to measure the global self-esteem of children and adolescent. The scale contains 10 items, which are rated on a 4-point Likert scale with score 1 to 4 (1= "strongly disagree", 2= "disagree", 3= "agree", 4 = "strongly agree"), with total possible scores ranging from 10 to 40. Higher scores indicate higher levels of self-esteem. Subjects will be asked to respond to the Chinese version of the RSES at baseline.
Change in level of self-esteem from baseline at 6-month between intervention and control group | 6-month follow-up
  The subjects' self-esteem will be assessed at 6-month follow-up, using the Chinese version of the Rosenberg Self-Esteem Scale (RSES).
  The RSES is a tool designed to measure the global self-esteem of children and adolescent. The scale contains 10 items, which are rated on a 4-point Likert scale with score 1 to 4 (1= "strongly disagree", 2= "disagree", 3= "agree", 4 = "strongly agree"), with total possible scores ranging from 10 to 40. Higher scores indicate higher levels of self-esteem. Subjects will be asked to respond to the Chinese version of the RSES at 6-month after starting the intervention.
Change in level of self-esteem from baseline at 12-month between intervention and control group | 12-month follow-up
  The subjects' self-esteem will be assessed at 12-month follow-up, using the Chinese version of the Rosenberg Self-Esteem Scale (RSES).
  The RSES is a tool designed to measure the global self-esteem of children and adolescent. The scale contains 10 items, which are rated on a 4-point Likert scale with score 1 to 4 (1= "strongly disagree", 2= "disagree", 3= "agree", 4 = "strongly agree"), with total possible scores ranging from 10 to 40. Higher scores indicate higher levels of self-esteem. Subjects will be asked to respond to the Chinese version of the RSES at 12-month after starting the intervention.
Quality of life at baseline between intervention and control group | baseline
  The subjects' quality of life will be assessed at baseline, using the Chinese version of the Paediatric Quality of Life Inventory 4.0 Generic Core Scale (PedsQL 4.0). The PedsQL is designed to measure children's health-related quality of life. The scale consists of 23 items which are categorized into four dimensions, namely physical functioning (8 items), emotional functioning (5 items), social functioning (5 items) and school functioning (5 items). All items are rated on a 5-point Likert scale from 0 (never) to 4 (almost always) by which the participants will be asked how much of a problem has been experienced over the last month. A total possible scores ranging from 0 to 100 will be obtained, with higher scores indicating better health-related quality of life. Subjects will be asked to respond to the Chinese version of the PedsQL 4.0 at baseline.
Change in Quality of life at 6-month follow-up between intervention and control group | 6-month follow-up
  The subjects' quality of life will be assessed at 6-month after starting the intervention, using the Chinese version of the Paediatric Quality of Life Inventory 4.0 Generic Core Scale (PedsQL 4.0). The PedsQL is designed to measure children's health-related quality of life. The scale consists of 23 items which are categorized into four dimensions, namely physical functioning (8 items), emotional functioning (5 items), social functioning (5 items) and school functioning (5 items). All items are rated on a 5-point Likert scale from 0 (never) to 4 (almost always) by which the participants will be asked how much of a problem has been experienced over the last month. A total possible scores ranging from 0 to 100 will be obtained, with higher scores indicating better health-related quality of life. Subjects will be asked to respond to the Chinese version of the PedsQL 4.0 at 6-month after starting the intervention.
Change in Quality of life at 12-month follow-up between intervention and control group | 12-month follow-up
  The subjects' quality of life will be assessed at 12-month after starting the intervention, using the Chinese version of the Paediatric Quality of Life Inventory 4.0 Generic Core Scale (PedsQL 4.0). The PedsQL is designed to measure children's health-related quality of life. The scale consists of 23 items which are categorized into four dimensions, namely physical functioning (8 items), emotional functioning (5 items), social functioning (5 items) and school functioning (5 items). All items are rated on a 5-point Likert scale from 0 (never) to 4 (almost always) by which the participants will be asked how much of a problem has been experienced over the last month. A total possible scores ranging from 0 to 100 will be obtained, with higher scores indicating better health-related quality of life. Subjects will be asked to respond to the Chinese version of the PedsQL 4.0 at 12-month after starting the intervention.

CONTACTS AND LOCATIONS:
Overall Officials: Ho Cheung William Li, Principal Investigator — The University of Hong Kong
Locations (1):
- The University of Hong Kong, Hong Kong, China

IPD SHARING:
Plan to Share IPD: No